CLINICAL TRIAL: NCT04580511
Title: Safety and Clinical Performance of a Non-cross-linked Porcine Acellular Dermal Matrix Used in Abdominal Wall Reconstruction: an Observational Prospective Study.
Brief Title: Safety and Clinical Performance of a Biological Matrix Used in Abdominal Wall Reconstruction
Acronym: PMCF_AWR
Status: Active, not recruiting | Type: Observational
Sponsor: Meccellis Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: AWR_01_CIP
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Wall Defect; Abdominal Wall Injury; Abdominal Hernia
Keywords: abdominal wall reconstruction; biological mesh
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CELLIS (Porcine Acellular Dermal Matrix, PADM) — Biological membrane used in abdominal reconstruction

SUMMARY:
The general objective of the study is to confirm the medium/long-term safety and clinical performance of the CELLIS membrane used in abdominal wall reconstruction including, but not limited to, ventral hernia repair and stoma closure, and to identify emerging risks in comparison to the clinical data related to other types of fixation material.

The present study will be a prospective multicentric non-randomized and noncontrolled trial involving 112 patients followed for 24 months. The study will be conducted in France in 3 investigational centres.

DETAILED DESCRIPTION:
The study will be prospective, multicentric, single-arm, observational (non-interventional) to evaluate the safety and performance of the CELLIS membrane used in abdominal wall reconstruction including, but not limited to, ventral hernia repair and stoma closure.

All evaluations will be performed and products used according to the usual practice, without additional or unusual diagnostic, treatment and monitoring procedure.

The study will be conducted in France in 3 investigational centres including 112 patients scheduled for an abdominal wall reconstruction.

Each patient will participate in one assessment period including a preoperative visit, followed by the day of surgical procedure and a hospitalization period.

Patients will return for ambulatory visits on day 30 (+/- 7 days), on month 3 (+/- 2 weeks), on month 12 (+/- 2 weeks) and on month 24 (+/-2 weeks) post-surgery.

CELLIS will be implanted by open technique following standard techniques. The membrane can be used in bridged or reinforced repairs. Mesh placement can include inlay (bridging), underlay intraperitoneal, sublay (retrorectus/retromuscular) positions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥18 years,
* Patient with an indication of abdominal wall reconstruction including, but not limited to, ventral hernia repair and stoma closure,
* Patient being informed of its participation to the study and of the follow-up visits, and having no objection to the clinical data collection and medical file access,
* Patient being informed of the porcine origin of the device in advance of the procedure.

Exclusion Criteria:

* Patient with known hypersensitivity to porcine materials,
* Patient who is pregnant,
* Patient having refused to participate to the study,
* Patient refusing to return for the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with an indication of abdominal wall reconstruction including, but not limited to, ventral hernia repair and stoma closure.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events including reoperation and removal of the mesh. The main complications of interest are Surgical Site Occurrence (SSO) including Surgical Site Infection (SSI). | From the surgical procedure throughout the entire 24-month follow-up period
  Percentage

SECONDARY OUTCOMES:
Rate of recurrence/incisional hernia evaluated by clinical examination and/or CT-scan | Throughout the study until end of the 24-month follow-up period
  Percentage
Rate of recurrence/incisional hernia requiring reoperation | Throughout the study until end of the 24-month follow-up period
  Percentage
Rate of abdominal wall laxity | Throughout the study until end of the 24-month follow-up period
  Percentage
Description of device deficiency: inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling. | During the surgical procedure
  Summarized and listed

CONTACTS AND LOCATIONS:
Overall Officials: Hassan BOUYABRINE, MD, Principal Investigator — CHU Montpellier, France
Locations (4):
- France (4):
  - CHU Caen Normandie, Service de Chirurgie Digestive, Caen
  - Groupe Hospitalier La Rochelle - Ré - Aunis, La Rochelle
  - CHU Montpellier, Hôpital Saint-Eloi, Pôle digestif, Service de Chirurgie Digestive B et Transplantation, Montpellier
  - CHU Nantes Hôtel Dieu, Nantes

IPD SHARING:
Plan to Share IPD: No